CLINICAL TRIAL: NCT06140992
Title: PaCIFiC-CUP：Pan-Cancer Integrated Fingerprinting Classifier for Identifying the Origin of Cancer of Unknown Primary: A Multi-Center Prospective Cohort Study
Brief Title: PaCIFiC-CUP Classifies Cancer of Unknown Primary
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Cancer Hospital (Other); Dongguan People's Hospital (Other Government); Beijing Tongren Hospital (Other); Anhui Provincial Hospital (Other Government); Peking University Third Hospital (Other); Henan Cancer Hospital (Other Government); Ganzhou Cancer Hospital (Unknown); Guangzhou Chest Hospital. (Unknown); First Affiliated Hospital of Jinan University (Other); Peking University Shenzhen Hospital (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiao-Peng Tian, Principal Investigator, Sun Yat-sen University
Other Study IDs: PaCIFiC-CUP
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Unknown Primary Tumors; DNA Methylation
Keywords: Unknown Primary Tumors; DNA methylation; Large Language Model; Pan-cancer
MeSH Terms: conditions — Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Site-Specific Therapy Group: These patients with cancer of unknown primary received site-specific therapy that matched the particular site predicted by the DNA methylation classifier.
- Empirical Therapy Group: These patients with cancer of unknown primary received empirical therapy that didn't match the particular site predicted by the DNA methylation classifier.

SUMMARY:
This study aims to initially utilize machine learning on pan-cancer DNA methylation data from public databases to construct a DNA methylation classification model (PaCIFiC-CUP, pan-cancer integrated fingerprinting classifier of CUP) for diagnosing various types of cancer, particularly the primary site of cancer of unknown primary. The goal is to achieve diagnosis of cancer pathology type by analyzing the DNA methylation patterns of cancer specimens, thereby guiding subsequent precision treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patient specimens were obtained from the Sun Yat-sen University Cancer Center and affiliated cooperating centers, with written consent from the patients authorizing the use of the specimens for research purposes.
2. Following standard assessments (medical history, physical examination, complete blood count, biochemistry, computed tomography scans of the neck, chest, abdomen, and pelvis, targeted evaluations of all symptomatic areas, pathology, and immunohistochemistry), the diagnosis was determined as a primary site unknown tumor (including adenocarcinoma, squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma, sarcoma, etc).
3. The diagnosis was confirmed at the participating institution and the patient had received systemic therapy.
4. Complete clinical, pathological, and follow-up data for the patients can be obtained.
5. ECOG performance status score: 0-2 points.

Exclusion Criteria:

1. Pregnant or lactating female patients.
2. Tumor tissue sample size is too small (tumor tissue accounts for <70% in the biopsy or slice tissue).
3. Organ transplant or history of non-autologous (allogeneic) bone marrow or stem cell transplantation.
4. History of previous tumors, with the current condition being a recurrent tumor.
5. Hematological malignancies (excluding lymphoma).
6. Other diseases that may severely impact patient survival, such as severe cardiovascular or cerebrovascular diseases, sepsis, severe trauma or burns, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with CUP who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of diagnosis until the date of death from any cause, assessed up to 24 months
  Overall survival refers to the length of time that a person lives after being diagnosed with cancer of unknown primary, without regard to any specific cause of death.

SECONDARY OUTCOMES:
Progression-Free Survival | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-Free Survival refers to the length of time during which a patient with cancer of unknown primary remains alive without any signs or symptoms of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramer A, Bochtler T, Pauli C, Baciarello G, Delorme S, Hemminki K, Mileshkin L, Moch H, Oien K, Olivier T, Patrikidou A, Wasan H, Zarkavelis G, Pentheroudakis G, Fizazi K; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Cancer of unknown primary: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Mar;34(3):228-246. doi: 10.1016/j.annonc.2022.11.013. Epub 2022 Dec 20. No abstract available. PMID 36563965
- [Background] Paziewska A, Dabrowska M, Goryca K, Antoniewicz A, Dobruch J, Mikula M, Jarosz D, Zapala L, Borowka A, Ostrowski J. DNA methylation status is more reliable than gene expression at detecting cancer in prostate biopsy. Br J Cancer. 2014 Aug 12;111(4):781-9. doi: 10.1038/bjc.2014.337. Epub 2014 Jun 17. PMID 24937670
- [Background] Wehmas LC, Hester SD, Wood CE. Direct formalin fixation induces widespread transcriptomic effects in archival tissue samples. Sci Rep. 2020 Sep 2;10(1):14497. doi: 10.1038/s41598-020-71521-w. PMID 32879405
- [Background] Capper D, Jones DTW, Sill M, Hovestadt V, Schrimpf D, Sturm D, Koelsche C, Sahm F, Chavez L, Reuss DE, Kratz A, Wefers AK, Huang K, Pajtler KW, Schweizer L, Stichel D, Olar A, Engel NW, Lindenberg K, Harter PN, Braczynski AK, Plate KH, Dohmen H, Garvalov BK, Coras R, Holsken A, Hewer E, Bewerunge-Hudler M, Schick M, Fischer R, Beschorner R, Schittenhelm J, Staszewski O, Wani K, Varlet P, Pages M, Temming P, Lohmann D, Selt F, Witt H, Milde T, Witt O, Aronica E, Giangaspero F, Rushing E, Scheurlen W, Geisenberger C, Rodriguez FJ, Becker A, Preusser M, Haberler C, Bjerkvig R, Cryan J, Farrell M, Deckert M, Hench J, Frank S, Serrano J, Kannan K, Tsirigos A, Bruck W, Hofer S, Brehmer S, Seiz-Rosenhagen M, Hanggi D, Hans V, Rozsnoki S, Hansford JR, Kohlhof P, Kristensen BW, Lechner M, Lopes B, Mawrin C, Ketter R, Kulozik A, Khatib Z, Heppner F, Koch A, Jouvet A, Keohane C, Muhleisen H, Mueller W, Pohl U, Prinz M, Benner A, Zapatka M, Gottardo NG, Driever PH, Kramm CM, Muller HL, Rutkowski S, von Hoff K, Fruhwald MC, Gnekow A, Fleischhack G, Tippelt S, Calaminus G, Monoranu CM, Perry A, Jones C, Jacques TS, Radlwimmer B, Gessi M, Pietsch T, Schramm J, Schackert G, Westphal M, Reifenberger G, Wesseling P, Weller M, Collins VP, Blumcke I, Bendszus M, Debus J, Huang A, Jabado N, Northcott PA, Paulus W, Gajjar A, Robinson GW, Taylor MD, Jaunmuktane Z, Ryzhova M, Platten M, Unterberg A, Wick W, Karajannis MA, Mittelbronn M, Acker T, Hartmann C, Aldape K, Schuller U, Buslei R, Lichter P, Kool M, Herold-Mende C, Ellison DW, Hasselblatt M, Snuderl M, Brandner S, Korshunov A, von Deimling A, Pfister SM. DNA methylation-based classification of central nervous system tumours. Nature. 2018 Mar 22;555(7697):469-474. doi: 10.1038/nature26000. Epub 2018 Mar 14. PMID 29539639
- [Background] Koelsche C, Schrimpf D, Stichel D, Sill M, Sahm F, Reuss DE, Blattner M, Worst B, Heilig CE, Beck K, Horak P, Kreutzfeldt S, Paff E, Stark S, Johann P, Selt F, Ecker J, Sturm D, Pajtler KW, Reinhardt A, Wefers AK, Sievers P, Ebrahimi A, Suwala A, Fernandez-Klett F, Casalini B, Korshunov A, Hovestadt V, Kommoss FKF, Kriegsmann M, Schick M, Bewerunge-Hudler M, Milde T, Witt O, Kulozik AE, Kool M, Romero-Perez L, Grunewald TGP, Kirchner T, Wick W, Platten M, Unterberg A, Uhl M, Abdollahi A, Debus J, Lehner B, Thomas C, Hasselblatt M, Paulus W, Hartmann C, Staszewski O, Prinz M, Hench J, Frank S, Versleijen-Jonkers YMH, Weidema ME, Mentzel T, Griewank K, de Alava E, Martin JD, Gastearena MAI, Chang KT, Low SYY, Cuevas-Bourdier A, Mittelbronn M, Mynarek M, Rutkowski S, Schuller U, Mautner VF, Schittenhelm J, Serrano J, Snuderl M, Buttner R, Klingebiel T, Buslei R, Gessler M, Wesseling P, Dinjens WNM, Brandner S, Jaunmuktane Z, Lyskjaer I, Schirmacher P, Stenzinger A, Brors B, Glimm H, Heining C, Tirado OM, Sainz-Jaspeado M, Mora J, Alonso J, Del Muro XG, Moran S, Esteller M, Benhamida JK, Ladanyi M, Wardelmann E, Antonescu C, Flanagan A, Dirksen U, Hohenberger P, Baumhoer D, Hartmann W, Vokuhl C, Flucke U, Petersen I, Mechtersheimer G, Capper D, Jones DTW, Frohling S, Pfister SM, von Deimling A. Sarcoma classification by DNA methylation profiling. Nat Commun. 2021 Jan 21;12(1):498. doi: 10.1038/s41467-020-20603-4. PMID 33479225
- [Background] Hovestadt V, Remke M, Kool M, Pietsch T, Northcott PA, Fischer R, Cavalli FM, Ramaswamy V, Zapatka M, Reifenberger G, Rutkowski S, Schick M, Bewerunge-Hudler M, Korshunov A, Lichter P, Taylor MD, Pfister SM, Jones DT. Robust molecular subgrouping and copy-number profiling of medulloblastoma from small amounts of archival tumour material using high-density DNA methylation arrays. Acta Neuropathol. 2013 Jun;125(6):913-6. doi: 10.1007/s00401-013-1126-5. Epub 2013 May 14. No abstract available. PMID 23670100
- [Background] Pajtler KW, Witt H, Sill M, Jones DT, Hovestadt V, Kratochwil F, Wani K, Tatevossian R, Punchihewa C, Johann P, Reimand J, Warnatz HJ, Ryzhova M, Mack S, Ramaswamy V, Capper D, Schweizer L, Sieber L, Wittmann A, Huang Z, van Sluis P, Volckmann R, Koster J, Versteeg R, Fults D, Toledano H, Avigad S, Hoffman LM, Donson AM, Foreman N, Hewer E, Zitterbart K, Gilbert M, Armstrong TS, Gupta N, Allen JC, Karajannis MA, Zagzag D, Hasselblatt M, Kulozik AE, Witt O, Collins VP, von Hoff K, Rutkowski S, Pietsch T, Bader G, Yaspo ML, von Deimling A, Lichter P, Taylor MD, Gilbertson R, Ellison DW, Aldape K, Korshunov A, Kool M, Pfister SM. Molecular Classification of Ependymal Tumors across All CNS Compartments, Histopathological Grades, and Age Groups. Cancer Cell. 2015 May 11;27(5):728-43. doi: 10.1016/j.ccell.2015.04.002. PMID 25965575
- [Background] Sturm D, Orr BA, Toprak UH, Hovestadt V, Jones DTW, Capper D, Sill M, Buchhalter I, Northcott PA, Leis I, Ryzhova M, Koelsche C, Pfaff E, Allen SJ, Balasubramanian G, Worst BC, Pajtler KW, Brabetz S, Johann PD, Sahm F, Reimand J, Mackay A, Carvalho DM, Remke M, Phillips JJ, Perry A, Cowdrey C, Drissi R, Fouladi M, Giangaspero F, Lastowska M, Grajkowska W, Scheurlen W, Pietsch T, Hagel C, Gojo J, Lotsch D, Berger W, Slavc I, Haberler C, Jouvet A, Holm S, Hofer S, Prinz M, Keohane C, Fried I, Mawrin C, Scheie D, Mobley BC, Schniederjan MJ, Santi M, Buccoliero AM, Dahiya S, Kramm CM, von Bueren AO, von Hoff K, Rutkowski S, Herold-Mende C, Fruhwald MC, Milde T, Hasselblatt M, Wesseling P, Rossler J, Schuller U, Ebinger M, Schittenhelm J, Frank S, Grobholz R, Vajtai I, Hans V, Schneppenheim R, Zitterbart K, Collins VP, Aronica E, Varlet P, Puget S, Dufour C, Grill J, Figarella-Branger D, Wolter M, Schuhmann MU, Shalaby T, Grotzer M, van Meter T, Monoranu CM, Felsberg J, Reifenberger G, Snuderl M, Forrester LA, Koster J, Versteeg R, Volckmann R, van Sluis P, Wolf S, Mikkelsen T, Gajjar A, Aldape K, Moore AS, Taylor MD, Jones C, Jabado N, Karajannis MA, Eils R, Schlesner M, Lichter P, von Deimling A, Pfister SM, Ellison DW, Korshunov A, Kool M. New Brain Tumor Entities Emerge from Molecular Classification of CNS-PNETs. Cell. 2016 Feb 25;164(5):1060-1072. doi: 10.1016/j.cell.2016.01.015. PMID 26919435
- [Background] Pisanic TR 2nd, Wang Y, Sun H, Considine M, Li L, Wang TH, Wang TL, Shih IM. Methylomic Landscapes of Ovarian Cancer Precursor Lesions. Clin Cancer Res. 2020 Dec 1;26(23):6310-6320. doi: 10.1158/1078-0432.CCR-20-0270. Epub 2020 Aug 17. PMID 32817081
- [Background] Muller D, Gyorffy B. DNA methylation-based diagnostic, prognostic, and predictive biomarkers in colorectal cancer. Biochim Biophys Acta Rev Cancer. 2022 May;1877(3):188722. doi: 10.1016/j.bbcan.2022.188722. Epub 2022 Mar 17. PMID 35307512
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Nunes SP, Moreira-Barbosa C, Salta S, Palma de Sousa S, Pousa I, Oliveira J, Soares M, Rego L, Dias T, Rodrigues J, Antunes L, Henrique R, Jeronimo C. Cell-Free DNA Methylation of Selected Genes Allows for Early Detection of the Major Cancers in Women. Cancers (Basel). 2018 Sep 26;10(10):357. doi: 10.3390/cancers10100357. PMID 30261643
- [Background] Moran S, Martinez-Cardus A, Sayols S, Musulen E, Balana C, Estival-Gonzalez A, Moutinho C, Heyn H, Diaz-Lagares A, de Moura MC, Stella GM, Comoglio PM, Ruiz-Miro M, Matias-Guiu X, Pazo-Cid R, Anton A, Lopez-Lopez R, Soler G, Longo F, Guerra I, Fernandez S, Assenov Y, Plass C, Morales R, Carles J, Bowtell D, Mileshkin L, Sia D, Tothill R, Tabernero J, Llovet JM, Esteller M. Epigenetic profiling to classify cancer of unknown primary: a multicentre, retrospective analysis. Lancet Oncol. 2016 Oct;17(10):1386-1395. doi: 10.1016/S1470-2045(16)30297-2. Epub 2016 Aug 27. PMID 27575023
- [Background] Zhang Z, Lu Y, Vosoughi S, Levy JJ, Christensen BC, Salas LA. HiTAIC: hierarchical tumor artificial intelligence classifier traces tissue of origin and tumor type in primary and metastasized tumors using DNA methylation. NAR Cancer. 2023 Apr 19;5(2):zcad017. doi: 10.1093/narcan/zcad017. eCollection 2023 Jun. PMID 37089814
- [Background] Greco FA, Lennington WJ, Spigel DR, Hainsworth JD. Molecular profiling diagnosis in unknown primary cancer: accuracy and ability to complement standard pathology. J Natl Cancer Inst. 2013 Jun 5;105(11):782-90. doi: 10.1093/jnci/djt099. Epub 2013 May 2. PMID 23641043
- [Background] Maros ME, Capper D, Jones DTW, Hovestadt V, von Deimling A, Pfister SM, Benner A, Zucknick M, Sill M. Machine learning workflows to estimate class probabilities for precision cancer diagnostics on DNA methylation microarray data. Nat Protoc. 2020 Feb;15(2):479-512. doi: 10.1038/s41596-019-0251-6. Epub 2020 Jan 13. PMID 31932775